CLINICAL TRIAL: NCT02519881
Title: This Clinical Trial Evaluated the Efficacy and Safety of a Modified Microfracture Using Collagen Compared to Those of a Simple Microfracture in Patients With Cartilage Defects in Their Ankles.
Brief Title: the Efficacy and Safety of a Modified Microfracture Using Collagen Compared to Those of a Simple Microfracture in Ankle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04CAR
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Defect of Articular Cartilage
Keywords: cartilage defect in ankle; microfracture; modified microfracture using collagen; collagen
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified microfracture using collagen (Experimental): modified microfracture using collagen (CartiFill) for cartilage defect of ankle
  Interventions: Procedure: Microfracture; Device: CartiFill
- microfracture (Active Comparator): simple microfracture for cartilage defect of ankle
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: Microfracture — simple microfracture of ankle
Device: CartiFill — add collagen when doing microfracture
  Arms: modified microfracture using collagen

SUMMARY:
This study was designed to evaluate the efficacy and safety of a modified microfracture using collagen, and to compare them with those of a simple microfracture in patients with cartilage defects in their ankles.

DETAILED DESCRIPTION:
This study was an open-trial study. Sixty subjects participated in it. The study was explained to the subjects and they voluntarily agreed to participate in it. Their eligibility to participate in the study was checked, and they were randomized either into the simple microfracture group or the modified microfracture group using collagen based on a randomization table. They were asked to follow the guidelines of the investigators during the study and to visit the hospital five times, including for screening. At each visit, the subjects underwent an examination with doctors and MRI to evaluate the efficacy of the procedure. (*If the subject began the first visit on the screening date, the total number of his or her visits was four.)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were 15 years old or older
2. Patients with cartilage defects in their ankle
3. Patients with misalignment of their tibia and talus, unstable ligament in their ankle, or bony defects in the lesions of their ankle, and/or who had been treated for alignment
4. Patients or their representative (for adults), or patients and their parent/guardian (for minors), who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

1. If patients or their families suffer from or have ever suffered from an autoimmune disease.
2. Patients who have ever suffered an anaphylactic reaction.
3. Patients who have ever suffered hypersensitivity to an implant.
4. Patients with a history of allergy to porcine or bovine protein.
5. Subjects with inflammatory arthritis, such as rheumatoid and gouty arthritis.
6. Subjects with autoimmune disease related arthritis.
7. Subjects who are pregnant and/or breast-feeding and/or plan a pregnancy.
8. Subjects with tumors.
9. Subjects who have undergone radiotherapy or chemotherapy within the last 2 years (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).
10. Subjects who are diabetic. (Exception: if the possibility of CartiFill™ treatment is confirmed with doctor's clinical decision, and/or patient's blood glucose level remains within the normal range and/or no other complications by diabetes mellitus.)
11. Subjects with infections, currently on treatment with antibiotics or antimicrobials (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).
12. Subjects under adrenocorticoid therapy (Exception: if the possibility of collagen treatment is confirmed with doctor's clinical decision).
13. Subjects with psychiatric disorders who are considered inappropriate to participate in this trial by the Principal Investigator.
14. Patients who have ever suffered contraindications of the used Fibrin sealant. (The major contraindications are as follows: patients with hypersensitivity to aprotinin and those treatments for severe brisk arterial or venous bleeding.)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
100mmVAS(visual analogue scale) score | 12 months after the surgery
  The VAS's were evaluated 12 months after the surgery on the affected ankle in the study and control groups.

SECONDARY OUTCOMES:
Change score of 100mmVAS(visual analogue scale) | Screening, 6, 12, and 24months after surgery
  The difference in the 100mmVAS on the affected ankle at the screening and after 12 months was compared in the study and control group, as were the differences in the 100mmVAS after 6, and 24 months.
Change of Satisfaction evaluation by patients | Screening, 6, 12, and 24months after surgery
  The improvements in the affected ankle before and 12 months after the surgery (and six and 24 months after the surgery) were compared in the study and control group.
Change of AOFAS(American orthopaedic foot & ankle society) Score | Screening, 6, 12, and 24months after surgery
  The difference in the AOFAS on the affected ankle at the screening and after 12 months was compared in the study and control group, as were the differences in the AOFAS after 6, and 24 months.
Change of Hannover Score | Screening, 6, 12, and 24months after surgery
  The difference in the Hannover Score on the affected ankle at the screening and after 12 months was compared in the study and control group, as were the differences in the Hannover Score after 6, and 24 months.
Change of Satisfaction evaluation by physician in charge | Screening, 6, 12, and 24months after surgery
  The improvements in the affected ankle before and 12 months after the surgery (and six and 24 months after the surgery) were compared in the study and control group.
Change results of Arthroscopy (ICRS(International Cartilage Repair Society)) | before and 24 months after the surgery
  The conditions of the affected ankle before and 24 months after the surgery were recorded and the ICRS's were evaluated in the study and control group.
  * Arthroscopy was performed in up to 10 subjects who signed the consent form.
the result of MRI(mMOCART) | 24 months after the surgery
  The conditions of the affected ankle 24 months after the surgery were recorded and the mMOCART were evaluated in the study and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soo Kim, MD, Principal Investigator — Eulji General Hospital; Young Hwan Kim, MD, Principal Investigator — Soon Chun Hyang University; Hyung Nyun Kim, MD, Principal Investigator — Hallym University Medical Center-Kangnam Sacred Heart Hospital
Locations (3):
- South Korea (3):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Eulji general Hospital, Seoul, Seoul
  - Hallym University Medical Center-Kangnam Sacred Heart Hospital, Seoul, Seoul

REFERENCES:
- [Derived] Lee YK, Young KW, Kim JS, Lee HS, Cho WJ, Kim HN. Arthroscopic microfracture with atelocollagen augmentation for osteochondral lesion of the talus: a multicenter randomized controlled trial. BMC Musculoskelet Disord. 2020 Nov 3;21(1):716. doi: 10.1186/s12891-020-03730-3. PMID 33143647